

## Royal Devon and Exeter NHS Foundation Trust

## Timing of Suture Removal to Reduce Scarring in Skin Surgery

## **Participant Consent Form**

IRAS ID: 303519 Participant Number: Initials: I confirm that I have read the patient information sheet, v3, dated 9th September 2021 for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. I agree to my General Practitioner being informed of my participation in the study. I agree to having photos taken of my skin lesion, which will be uploaded directly to my electronic patient record I agree to my medical records being accessed by the research team for routinely collected data such as age, past medical history and surgical procedure notes I agree to take part in the above study. Participant: Date: ...../..... Signature: Name (please print): Consenter: Date: ...../...../ Signature: Name: (please print):